CLINICAL TRIAL: NCT02347046
Title: Clinical Pharmacology Study of FYU-981 for Subjects With Renal Insufficiency.
Brief Title: Clinical Pharmacology of FYU-981 (Subjects With Renal Insufficiency)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fuji Yakuhin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: FYU-981-005
Record Dates: First submitted 2015-01-16; First posted 2015-01-27 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-01

CONDITIONS: Renal Insufficiency; Healthy
MeSH Terms: conditions — Renal Insufficiency | interventions — dotinurad

ARMS (3):
- Moderately-decreased group (Experimental): (eGFR: >=30mL/min/1.73m^2 and < 60mL/min/1.73m^2)
  Interventions: Drug: FYU-981, (Oral single dosing)
- Slightly-decreased group (Experimental): (eGFR: >=60mL/min/1.73m^2 and < 90mL/min/1.73m^2)
  Interventions: Drug: FYU-981, (Oral single dosing)
- Normal group (Experimental): (eGFR: >=90mL/min/1.73m^2)
  Interventions: Drug: FYU-981, (Oral single dosing)

INTERVENTIONS:
Drug: FYU-981, (Oral single dosing) — FYU-981, (Oral single dosing)

SUMMARY:
The purpose of this study is to assess the pharmacokinetics, pharmacodynamics and safety after single oral administration of FYU-981 to subjects with renal insufficiency and with normal renal function.

ELIGIBILITY:
Inclusion Criteria:

* Japanese adult subjects
* Body mass index: >=18.5 and <30.0

Exclusion Criteria:

* Subjects with any disease or any history of diseases that might be unsuitable for participation in the clinical study

Min Age: 20 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (Cmax: Maximum plasma concentration) | 48 hours
Pharmacokinetics (Tmax: Time to reach the peak plasma concentration) | 48 hours
Pharmacokinetics (T1/2: Elimination half-life of plasma concentration) | 48 hours
Pharmacokinetics (AUC: Area under the plasma concentration-time curve) | 48 hours
Pharmacokinetics (CLtot/F: Total clearance / Fraction of dose absorbed) | 48 hours
Pharmacokinetics (kel: Elimination rate constant) | 48 hours
Pharmacokinetics (Vd/F: Distribution volume / Fraction of dose absorbed) | 48 hours
Pharmacokinetics (MRT: Mean residence time) | 48 hours
Pharmacokinetics (Ae: Amount of drug excreted in urine) | 48 hours
Pharmacokinetics (fe: Fraction of dose excreted in urine) | 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Japan, Kagoshima, Japan

REFERENCES:
- [Derived] Fukase H, Okui D, Sasaki T, Fushimi M, Ohashi T, Hosoya T. Effects of mild and moderate renal dysfunction on pharmacokinetics, pharmacodynamics, and safety of dotinurad: a novel selective urate reabsorption inhibitor. Clin Exp Nephrol. 2020 Mar;24(Suppl 1):17-24. doi: 10.1007/s10157-019-01825-3. Epub 2019 Dec 10. PMID 31823130